CLINICAL TRIAL: NCT03125473
Title: A Phase 1b, Open-Label, Dose-Optimization Trial of an Adenoviral-vector Based Norovirus Vaccine (VXA-G1.1-NN) Expressing GI.1 VP1 and dsRNA Adjuvant Administered Orally to Healthy Volunteers
Brief Title: Dose-Optimization Trial of VXA-G1.1-NN in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vaxart (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VXA-G11-102
Record Dates: First submitted 2017-04-14; First posted 2017-04-24 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Norovirus Gastroenteritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Group 1 (Experimental): Multiple doses of low dose VXA-G1.1-NN Oral Vaccine Tablets will be orally administered. VXA-G1.1-NN is an E1/E3-deleted replication-defective Adenovirus serotype 5 vaccine vector for prevention of noroviral gastroenteritis caused by Norovirus GI.1. The vaccine vector encodes for a full length VP1 (major capsid protein) gene from Norvirus GI.1 Norwalk. Subjects will receive 1 tablet of VXA-G1.1-NN on Days 1 and 8
  Interventions: Biological: VXA-G1.1-NN Oral Vaccine
- Dose Group 2 (Experimental): Multiple doses of low doseVXA-G1.1-NN Oral Vaccine Tablets will be orally administered. VXA-G1.1-NN is an E1/E3-deleted replication-defective Adenovirus serotype 5 vaccine vector for prevention of noroviral gastroenteritis caused by Norovirus GI.1. The vaccine vector encodes for a full length VP1 (major capsid protein) gene from Norvirus GI.1 Norwalk. Subjects will receive 1 tablet of VXA-G1.1-NN on Days 1, 3, and 5
  Interventions: Biological: VXA-G1.1-NN Oral Vaccine
- Dose Group 3 (Experimental): Multiple doses of low dose VXA-G1.1-NN Oral Vaccine Tablets will be orally administered. VXA-G1.1-NN is an E1/E3-deleted replication-defective Adenovirus serotype 5 vaccine vector for prevention of noroviral gastroenteritis caused by Norovirus GI.1. The vaccine vector encodes for a full length VP1 (major capsid protein) gene from Norvirus GI.1 Norwalk. Subjects will receive 1 tablet of VXA-G1.1-NN on Days 1 and 29.
  Interventions: Biological: VXA-G1.1-NN Oral Vaccine
- Dose Group 4 (Experimental): Multiple doses of low dose VXA-G1.1-NN Oral Vaccine Tablets will be orally administered. VXA-G1.1-NN is an E1/E3-deleted replication-defective Adenovirus serotype 5 vaccine vector for prevention of noroviral gastroenteritis caused by Norovirus GI.1. The vaccine vector encodes for a full length VP1 (major capsid protein) gene from Norvirus GI.1 Norwalk. Subjects will receive 6 tablets of VXA-G1.1-NN on Days 1 and 29
  Interventions: Biological: VXA-G1.1-NN Oral Vaccine

INTERVENTIONS:
Biological: VXA-G1.1-NN Oral Vaccine — The drug product will be provided as small white enteric-coated tablets. Multiple tablets will be administered to deliver the high total doses.
  Other Names: Active VXA-G.1.1-NN Oral Tablet Vaccine

SUMMARY:
A Phase 1b, randomized, double-blind, dose-ranging trial to determine the safety of different dosing regimens an adenoviral-vector based norovirus vaccine (VXA-G1.1-NN) expressing GI.1 VP1 and dsRNA adjuvant administered orally to healthy volunteers

DETAILED DESCRIPTION:
This study will enroll approximately 60 subjects in four cohorts of 15 subjects each. The cohorts may be enrolled and run in parallel or overlap; they do not have to run sequentially. The dosing for each cohort will be as follows:

Cohort 1: Multiple low dose on Days 1 and 8 Cohort 2: Multiple low dose on Days 1, 3 and 5 Cohort 3: Multiple low dose on Days 1 and 29 Cohort 4: Multiple high dose on Days 1 and 29

All subjects receiving study drug will have safety and immunogenicity assessments completed through Study Day 57 following their initial vaccination. Subjects may also be evaluated for persistent immunogenicity at Day 180 and will be followed for safety for 12 months following initial vaccination (Study Day 365).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female volunteers aged 19 - 49 years
2. Able to give written informed consent.
3. Healthy (no clinically significant health concerns), as determined by medical history, physical examination, 12-lead ECG, and vital signs at screening.
4. Safety laboratory values within the following range criteria at screening or abnormal and not clinically significant as outlined within the clinical protocol
5. Body mass index between 17 and 35 inclusively (kg/m2)
6. Comprehension of the study requirements with ability and willingness to complete all assessments and comply with scheduled visits and contacts.
7. Female participants must have a negative pregnancy test at baseline and fulfill one of the following criteria:

   1. At least one year post-menopausal;
   2. Surgically sterile;
   3. Willing to use oral, implantable, transdermal or injectable contraceptives for 30 days prior to and until 60 days after vaccination;
   4. A reliable form of contraception must be approved by the Investigator

Exclusion Criteria:

1. Receipt of any investigational norovirus vaccine within past 2 years
2. Administration of any investigational vaccine, drug or device within 8 weeks preceding vaccination, or planned use of the above stated during the study through the 12-month safety follow-up.
3. Administration of any licensed vaccine within 30 days prior to vaccination.
4. Presence of significant uncontrolled medical or psychiatric illness (acute or chronic) including institution of new medical/surgical treatment or dose alteration for uncontrolled symptoms or drug toxicity within 3 months
5. Any one of the following ECG findings within 30 days prior to vaccination:

   * QTcF interval duration > 460 msec (male) or > 470 msec (female),
   * QRS interval greater than 120 msec,
   * PR interval greater than 220 msec,
   * Clinically significant ST-T wave changes or pathologic Q waves.
6. Positive serology for HIV-1 or HIV-2, or HBsAg or HCV antibodies.
7. Cancer, or treatment for cancer treatment, within past 3 years (excluding history of basal cell carcinoma, squamous cell carcinoma, or cervical cancer in situ).
8. History of a hypersensitivity or allergic reaction to any component of the investigational vaccine or placebo, including but not limited to fish gelatin. Subjects with known fish allergies should be excluded.
9. Presence of immunosuppression or medical condition possibly associated with impaired immune responsiveness, including diabetes mellitus.
10. Administration of any medications or treatments that may adversely affect the immune system such as allergy injections, immune globulin, interferon, immunomodulators, cytotoxic drugs or other drugs known to be associated with significant major organ toxicity, or systemic corticosteroids (oral or injectable) during 3 months prior to vaccination. Inhaled and topical corticosteroids allowed.
11. Presence of household members who have received the Ad4 or Ad7 vaccines within 2 months prior to vaccination.
12. Presence of household members who are neonates, pregnant women, or hematopoietic stem cell transplant or solid organ transplant recipients from screening until the end of the active period
13. History of drug, alcohol or chemical abuse within 1 year prior to vaccination.
14. Receipt of blood or blood products 6 months prior to vaccination or planned administration during the follow-up study period.
15. Donation of blood or blood products within 4 weeks prior to vaccination or planned donation during the study period.
16. Acute disease within 72 hours prior to vaccination defined as the presence of a moderate or severe illness with or without fever.

    during screening period).
17. Presence of fever ≥38oC
18. Stool sample with occult blood
19. Positive urine drug screen for drugs of abuse
20. Positive urine alcohol test at
21. Consistent/habitual smoking within 2 months prior to vaccination.
22. History of serious reactions to any vaccination such as anaphylaxis, respiratory problems, hives or abdominal pain.
23. Diagnosed bleeding disorder or significant bruising or bleeding difficulties that could make blood draws problematic.
24. History of irritable bowel disease or other inflammatory digestive or gastrointestinal condition that could affect the distribution / safety evaluation of an orally administered vaccine targeting the mucosa of the small intestine.

Ages: 19 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2017-04-07 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2018-05-06 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety of different dosing regimens of VXA-G1.1-NN vaccine as determined by the incidence of treatment-emergent adverse events, physical exams, vital signs, and clinical laboratory test results (hematology, serum chemistry, and urinalysis). | Day 1 thru Day 57
  Safety will be evaluated by local and systemic reactogenicity (solicited symptoms), and clinical and laboratory assessments including physical exams, vital signs, clinical laboratory tests (hematology, serum chemistry, and urinalysis), and adverse events (AEs).

SECONDARY OUTCOMES:
Evaluate the effect of different dosing regimens of VXA-G1.1-NN vaccine on its immunogenicity as determined by cellular and humoral immune function assays performed on blood samples collected at preselected study visits. | Day 1 thru Day 180
  All subjects will have blood samples collected on study days 7, 28, and 57 following their initial vaccination for cellular and humoral immune function assays (i.e., production of vaccine specific blocking and neutralizing antibodies, formation of vaccine specific antibody secreting and memory cells, etc.) to assess the effect of the different dosing schedules on the immunogenicity of the VXA-G1.1-NN vaccine. Subjects may also be evaluated for persistent immunogenicity at Day 180 (optional).

CONTACTS AND LOCATIONS:
Overall Officials: Laura Sterling, MD, Principal Investigator — Celerion
Locations (1):
- Celerion, Inc., Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Undecided